CLINICAL TRIAL: NCT00125151
Title: Pharmacokinetics, Clinical Efficacy and Safety of C1 Inhibitor Concentrate (C1-Esteraseremmer-N) for the Treatment of Hereditary (and Acquired) Angioedema
Brief Title: C1-Esteraseremmer-N for the Treatment of Hereditary (and Acquired) Angioedema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prothya Biosolutions (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KB2003.01B
Record Dates: First submitted 2005-07-28; First posted 2005-07-29 (Estimated); Last update posted 2009-05-04 (Estimated); Status verified 2009-05

CONDITIONS: Angioedema
Keywords: MeSH: angioneurotic edema, complement 1 inactivators; Hereditary angioedema type I or II, Acquired angioedema
MeSH Terms: conditions — Angioedema; Hereditary Angioedema Types I and II; Acquired angioedema

INTERVENTIONS:
Drug: C1 inhibitor concentrate (C1-esteraseremmer-N)

SUMMARY:
A multicentre study to investigate the pharmacokinetics, clinical efficacy and safety of nanofiltered Cetor® (called C1-esteraseremmer-N during the development phase) for the treatment of hereditary angioedema (HAE) will be performed. This study (KB2003.01) consists of three parts: Part A - pharmacokinetics (phase II); Part B - treatment of attacks of angioedema (phase III); and Part C - prophylactic use of C1 inhibitor (phase III). Parts B + C will provide data on the efficacy of C1-esteraseremmer-N.

The changes within the manufacturing process of C1-esteraseremmer-N, compared to Cetor® nanofiltration and omission of hepatitis B immunoglobulin, most likely will not affect tolerability. The nanofiltration will provide more safety regarding viruses.

In Part B of the study, 15 attacks of hereditary angioedema will be treated with open-label C1-esteraseremmer-N. Attack severity and duration will be monitored by the subjective experience of the patient himself (which has been shown to be the most sensitive way of monitoring attack severity) and compared with historical (and literature) data. If possible, some attacks of acquired angioedema will also be included.

DETAILED DESCRIPTION:
A multicentre study to investigate the pharmacokinetics, clinical efficacy and safety of nanofiltered Cetor® (called C1-esteraseremmer-N during the development phase) for the treatment of hereditary angioedema (HAE) will be performed. This study (KB2003.01) consists of three parts: Part A - pharmacokinetics (phase II); Part B - treatment of attacks of angioedema (phase III); and Part C - prophylactic use of C1 inhibitor (phase III). Parts B + C will provide data on the efficacy of C1-esteraseremmer-N.

The changes within the manufacturing process of C1-esteraseremmer-N, compared to Cetor® nanofiltration and omission of hepatitis B immunoglobulin, most likely will not affect tolerability. The nanofiltration will provide more safety regarding viruses.

In Part B of the study, 15 attacks of hereditary angioedema will be treated with open-label C1-esteraseremmer-N. Attack severity and duration will be monitored by the subjective experience of the patient himself (which has been shown to be the most sensitive way of monitoring attack severity) and compared with historical (and literature) data. If possible, some attacks of acquired angioedema will also be included.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for HAE type I and type II patients:

* Established diagnosis of hereditary angioedema (type I or II): markedly decreased C1 inhibitor activity; decreased (type I), normal or elevated (type II) level of C1 inhibitor antigen; decreased level of C4.
* Age ≥ 16 years
* Evidence of a peripheral, abdominal, facial, laryngeal or genitourinary attack of angioedema of moderate to severe intensity, starting less then 5 hours before infusion. An attack is defined as moderate if it affects the normal daily activities of the patient in any way. Severe attacks are defined by the inability to perform normal daily activities.
* Signed informed consent by patient and patient's legal representative if under 18 years old

Inclusion criteria for acquired angioedema patients:

* Established diagnosis of acquired angioedema: recurrent attacks of angioedema without urticaria; no family history; decreased functional C1 inhibitor; decreased level of C4.
* Autoantibodies to C1 inhibitor or decreased C1q or onset after the third decade of life.
* Age ≥ 16 years
* Evidence of a peripheral, abdominal, facial, laryngeal or genitourinary attack of angioedema of moderate to severe intensity, starting less then 5 hours before infusion. An attack is defined as moderate if it affects the normal daily activities of the patient in any way. Severe attacks are defined by the inability to perform normal daily activities.
* Currently treated with C1 inhibitor concentrate to reverse angioedema.
* Signed informed consent by patient and patient's legal representative if under 18 years old

Exclusion Criteria:

Exclusion criteria for HAE type I and type II patients:

* Presence of clinically-relevant anti-C1 inhibitor auto-antibodies
* Participation in another pharmaceutical clinical study, which can interfere with this study, in the last 3 months prior to the study, other than Part A of this protocol.
* Addiction to narcotic/pain medication in case of an abdominal attack
* B-cell malignancy
* Use of narcotic medication within 3 days prior to attack.
* Use of heparin within the last two days prior to the study
* Pregnancy or lactation
* History of allergic reactions to C1 inhibitor concentrate or other blood products

Exclusion criteria for acquired angioedema patients:

* Participation in another pharmaceutical clinical study, which can interfere with this study, in the last 3 months prior to the study
* Addiction to narcotic/pain medication in case of an abdominal attack
* Use of narcotic medication within 3 days prior to attack.
* Use of heparin within the last two days prior to the study
* Pregnancy or lactation.
* History of allergic reactions to C1 inhibitor concentrate or other blood products

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2006-02; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
The primary objective in this clinical study, in which patients use C1-esteraseremmer-N to treat an attack of angioedema, is to investigate the efficacy and the time-to-effect of C1-esteraseremmer-N.

SECONDARY OUTCOMES:
Secondary objectives are the safety of C1-esteraseremmer-N and the ability of C1-esteraseremmer-N to increase the C1 inhibitor level and activity.

CONTACTS AND LOCATIONS:
Overall Officials: M. M. Levi, Prof. Dr., Principal Investigator — Academic Medical Centre Amsterdam
Locations (3):
- Netherlands (3):
  - Academic Medical Centre, Amsterdam
  - Academic hospital Groningen, Groningen
  - Erasmus Medical Centre, Rotterdam